CLINICAL TRIAL: NCT05726370
Title: A Phase 2 Study of Preoperative Pembrolizumab and Chemotherapy Followed by Adjuvant Pembrolizumab in Resectable Locoregionally Recurrent Head and Neck Squamous Cell Carcinoma
Brief Title: Preoperative Pembrolizumab and Chemotherapy in Resectable, Recurrent HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kartik Sehgal, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-504
Record Dates: First submitted 2023-01-24; First posted 2023-02-13 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Head and Neck Cancer; Resectable Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Second Primary Squamous Cell Carcinoma of the Head and Neck
Keywords: Head and Neck Squamous Cell Carcinoma; Head and Neck Cancer; Resectable Head and Neck Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Second Primary Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — pembrolizumab; Cisplatin; Carboplatin; Docetaxel; Taxoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pre-Operative Treatment + Salvage Surgery + Adjuvant Treatment (Experimental): Participants will complete study procedures as outlined:
  Preoperative Phase:
  * Mandatory biopsy at baseline.
  * Neoadjuvant treatment (2 cycles):
    * Cycles 1 - 2 ---Day 1 of 21-day Cycle: Predetermined doses of Pembrolizumab, Cisplatin (or Carboplatin) and Docetaxel.
  Surgery:
  -Primary tumor resection and/or lymph node dissection surgery 3-6 weeks from cycle 2 day 1
  Adjuvant Phase:
  -3-8 weeks post-surgery and upto a total of 15 cycles
  --Cycles 3 - 17
  ---Day 1 of 21-day cycle: Predetermined dose of Pembrolizumab
  Follow up appointments
  Interventions: Drug: Pembrolizumab; Drug: CISPLATIN; Drug: Carboplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Pembrolizumab — Immunoglobulin G4 monoclonal antibody, via IV infusion
  Other Names: MK-3475
Drug: CISPLATIN — Platinum agent, via IV infusion
Drug: Carboplatin — Platinum agent, via IV infusion
Drug: Docetaxel — Antineoplastic agent, via IV infusion.
  Other Names: Taxanes

SUMMARY:
This research study is evaluating effectiveness and safety of a combination of immunotherapy drug, pembrolizumab, with chemotherapy, as a possible treatment before and after surgery for squamous cell carcinoma of the head and neck (HNSCC). The combination of pembrolizumab and chemotherapy will be given prior to your surgery, while immunotherapy pembrolizumab will be continued for approximately 1 year after surgery.

The names of the study drugs involved in this research study are:

* pembrolizumab (a type of immunotherapy)
* docetaxel (a type of chemotherapy)
* cisplatin (a type of chemotherapy)
* carboplatin (a type of chemotherapy)

DETAILED DESCRIPTION:
This is a Phase II, open-label, non-randomized, single arm, single-center interventional study of neoadjuvant chemoimmunotherapy with pembrolizumab, cisplatin (or carboplatin), and docetaxel followed by surgery followed by adjuvant pembrolizumab therapy in patients with resectable recurrent squamous cell carcinoma of the head and neck (HNSCC). This study will also include individuals with new HNSCC which developed in a field that has received prior radiation therapy. Pembrolizumab works by helping the immune system to fight HNSCC.

This research study involves screening for eligibility, study treatment visits including evaluations, radiologic scans, tumor biopsies, and blood tests.

The U.S. Food and Drug Administration (FDA) has not approved Pembrolizumab for squamous cell carcinoma of the head and neck (HNSCC) setting before and after surgery, but it has been approved for HNSCC in the advanced incurable setting when surgery is no longer possible or cancer has spread to parts of the body outside the head and neck region.

All other drugs used in this study have been approved by the FDA for squamous cell carcinoma of the head and neck (HNSCC) in the advanced incurable setting.

Participation in this research study is expected to last for up to 5 years.

It is expected that about 28 people will take part in this research study.

Merck Sharp & Dohme LLC is supporting this research study and providing the study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed locoregionally recurrent squamous cell carcinoma of the head and neck, or second primary HNSCC in a previously irradiated field, defined as >50% of the presurgical tumor volume having prior radiation dose of >45 Gy as determined by the treating radiation oncologist (including primary sites, such as oral cavity, oropharynx, larynx or hypopharynx carcinoma).
* Participants must be a candidate for curative intent surgery.
* Participants must have documented time of ≥ 6 months from completion of prior curative intent treatment for HNSCC (surgery and/or radiation therapy with/without platinum chemotherapy or cetuximab targeted therapy) to diagnosis of local or locoregional recurrence or a second primary in a previously irradiated field.
* Participants must be willing to undergo a mandatory pre-treatment biopsy and willing to provide blood and tissue from the pre-treatment biopsy and at the time of surgery. Exceptions may be made after discussion with sponsor if it is not medically feasible to obtain a pre-treatment biopsy or is in the best interest of the patient. Archival tissue may be collected in this situation. Participants will be offered the opportunity to volunteer for optional biopsies at the time of recurrence of disease.
* Participants may have any smoking history (no restrictions)
* Participants may have any Human Papilloma Virus (HPV) status of the tumor. Patients with oropharyngeal cancer are required to undergo HPV testing with p16 immunohistochemistry and/or confirmatory HPV PCR or ISH testing
* Age ≥18 years
* ECOG performance status 0 or 1 (Karnofsky ≥70%, see Appendix A)
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes ≥3,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * total bilirubin ≤ institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN
  * creatinine ≤ institutional ULN OR
  * glomerular filtration rate (GFR) ≥50 mL/min/1.73 m2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m2.
* Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Because pembrolizumab and chemotherapy can be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Male participants: A male participant must agree to use a contraception as detailed in Appendix B of this protocol during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.
* Female participants: A female participant is eligible to participate if she is not pregnant (see Appendix B), not breastfeeding, and at least one of the following conditions applies:

  * a. Not a woman of childbearing potential (WOCBP) as defined in Appendix B OR
  * b. A WOCBP who agrees to follow the contraceptive guidance in Appendix B during the treatment period and for at least 180 days after the last dose of study treatment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Sinonasal, nasopharyngeal or cutaneous primary site of squamous cell carcinoma of the head and neck
* Has known distant metastatic disease. Those with known brain metastases should be excluded from this clinical trial, because of the poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, baseline brain imaging is not required prior to enrollment in the study if patients are asymptomatic
* Has had chemotherapy or radiotherapy for HNSCC in curative intent setting within 6 months prior to entering the study.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has a known additional malignancy that is progressing or has required active treatment within the past 2 years. Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (eg, breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
* Has a history of allergic reactions to agents used in study
* Has active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection. No HIV testing is required unless mandated by local health authority
* Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Has not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 2) with the exception of alopecia
* Has had an allogeneic tissue/solid organ transplant
* A WOCBP who has a positive urine pregnancy test within 72 hours prior to study registration (see Appendix B). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Pregnant women are excluded from this study because pembrolizumab and chemotherapy agents have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab and chemotherapy, breastfeeding should be discontinued if the mother is treated on this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-05-20 (Estimated)

PRIMARY OUTCOMES:
Rate of Major Pathological Response (mPR) | 2 months
  Major pathologic response (mPR) is defined as having ≤ 10% invasive squamous cell carcinoma within the resected primary tumor specimen and all sampled regional lymph nodes as assessed by pathologists. Rate is the proportion of treated participants who experienced mPR.

SECONDARY OUTCOMES:
Grade 3-5 Treatment-related Toxicity Rate | Up to 18 months
  Rate is the proportion of treated participants experiencing at least one treatment-related grade 3-5 AE of any type during the time of observation. All grade 3-5 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv5 as reported on case report forms were counted.
Median Overall Survival (OS) | Every six months up to 5 years
  OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Median Disease-Free Survival (DFS) | Every six months up to 5 years
  Disease-Free Survival (DFS) based on the Kaplan-Meier method is defined as the time from surgery to the first recurrence or death from any cause, whichever occurs first. Participants alive without disease recurrence are censored at date of last disease evaluation.
Best Radiological Response Rate | Before Salvage Surgery, upto 10 weeks from study registration
  Best radiological response are based on the RECIST 1.1 criteria, defined protocol section 11.2.4.

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Sehgal, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu